CLINICAL TRIAL: NCT02519660
Title: Lidocaine/Tetracaine Patch (Ralydan) vs Lidocaine/Prilocaine Cream (EMLA) for Needle Related Procedures in Children: a Multicenter, Randomized Controlled Trial
Brief Title: Needle Procedures Success Rate After Application of Ralydan vs EMLA in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 6/13
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Procedural Pain Relief
Keywords: Ralydan; EMLA cream; Procedural pain; Phlebotomy; Child
MeSH Terms: conditions — Pain, Procedural | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine/Tetracaine patch (Ralydan) (Experimental): Ralydan patch is a drug delivery system designed to release local anaesthetics (lidocaine and tetracaine) through the skin. It is applied in the site of venipuncture 30 minutes before needle procedure
  Interventions: Drug: Lidocaine/Tetracaine patch
- Lidocaine/Prilocaine cream (EMLA) (Active Comparator): EMLA cream is an eutectic mixture of local anaesthetic (lidocaine, prilocaine). It is applied in the site of venipuncture 60 minutes before needle procedure
  Interventions: Drug: Lidocaine/Prilocaine cream

INTERVENTIONS:
Drug: Lidocaine/Tetracaine patch
  Other Names: Ralydan
  Arms: Lidocaine/Tetracaine patch (Ralydan)
Drug: Lidocaine/Prilocaine cream
  Other Names: EMLA
  Arms: Lidocaine/Prilocaine cream (EMLA)

SUMMARY:
Needle-related procedures are among the most common sources of pain and distress for children in the health care setting. More than 50% of children reported pain during these procedures. The necessity for pain management during these procedures is well established. Topical anesthesia has been shown to be effective in managing needle-related pain. Eutectic mixture of local anaesthetic (EMLA) cream is the topical anesthetic most used. The application of this mixture of lidocaine and prilocaine reduce pain during needle procedures in children. To be effective EMLA cream must be applied for at least 60 minutes before needle procedure. This is the major limitation for its use in emergency settings.

Ralydan patch is a drug delivery system designed to release local anaesthetics (lidocaine and tetracaine) through the skin. There is evidence of pain relief after 30 minutes from its application. Only one randomized controlled trial compared the two topical anaesthetics in children during venipuncture and showed that Ralydan patch led to superior analgesia than EMLA cream, even if in this study the two anaesthetics were applied only for 35 minutes before needle procedure. No differences were found in success rate of the procedure and vein visibility. In adult patients, Ralydan and EMLA were equally effective in pain relief after 60 minutes from application.

To the best of the investigators' knowledge there is no published study that compared needle procedure success rate in children and pain relief effectiveness of lidocaine/tetracaine patch and lidocaine/prilocaine cream, at time of their maximum analgesic effect.

The aim of this study is to compare Ralydan patch and EMLA cream at time of their maximum analgesic effect (30 minutes vs 60 minutes), regard to needle procedure success rate at the first attempt and pain relief in children.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 10 years
* Need for peripheral IV line or venipuncture
* Informed consent signed by parents or legal guardians

Exclusion Criteria:

* Need for emergency care
* Known allergy or sensitivity to local anesthetics

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 339 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Success at the first attempt | Intraoperative
  Percentage of success at first attempt

SECONDARY OUTCOMES:
Pain score | Intraoperative
  The pain during the procedure will be evaluate using pain rating scale appropriate for age
Adverse events | Up to 15 minutes after the procedure
  The number and the type of adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Elena Neri, MD, Study Director — IRCCS Burlo Garofolo, Trieste, Italy; Giorgio Cozzi, MD, Principal Investigator — IRCCS Burlo Garofolo, Trieste, Italy
Locations (3):
- Italy (3):
  - Ospedale Pediatrico Pausilipon - Servizio di terapia del dolore e cure palliative, Napoli, Campania
  - IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia
  - Università degli studi di Padova - Centro Regionale Veneto di terapia del dolore e cure palliative pediatriche, Padua, Veneto